CLINICAL TRIAL: NCT02441231
Title: Probiotic Visbiome for Inflammation and Translocation in HIV II (PROOV IT II)
Brief Title: Probiotic Visbiome for Inflammation and Translocation in HIV II
Acronym: PROOV IT II
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: CIHR Canadian HIV Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTNPT 022B
Record Dates: First submitted 2015-04-23; First posted 2015-05-12 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic Group (Experimental): Visbiome probiotic group (900 billion bacteria daily; 2 sachets daily)
  Interventions: Drug: Visbiome
- Placebo Group (Placebo Comparator): Placebo comparator group
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Visbiome — Visbiome probiotic
  Arms: Probiotic Group
Other: Placebo — Placebo
  Arms: Placebo Group

SUMMARY:
Modern antiretroviral therapy (ART) has transformed the clinical care and lived experience of HIV infection. However, increased rates of adverse health conditions that are related to immune activation, such as cardiovascular disease (CVD) and neurodegenerative disease in ART-treated individuals persist. An important cause of this inflammation is the gut CD4 T cell loss and the "leaking" or translocation of luminal gut bacteria and other microbes across the bowel wall and into the bloodstream.

The use of complementary and alternative therapies is very common among people living with HIV, with estimates ranging from 16-60%. However, their efficacy has generally not been well demonstrated. Probiotics are live microbes that may provide a health benefit to the host and the investigators believe that the simultaneous use of probiotics along with ART will improve gut CD4 T cell restoration and function and therefore reduce microbial translocation and immune activation.

A major challenge to HIV treatment is the suboptimal CD4 T cell count despite successful HIV suppression on ART in immunologic non-responders (INRs). These individuals are at increased risk of AIDS-related deaths and non-AIDS related comorbidities that may be associated with increased immune activation and microbial translocation from the gut mucosa. With limited treatment options, alternative therapies to reduce inflammation and restore gut immunology will be important. Probiotic Visbiome consists of a high potency blend of eight different probiotics. The precise mechanism of action of Visbiome is unknown,but preclinical studies have shown that Visbiome may modulate the immune response towards an immunoregualtory phenotype with increased the levels of IL-10 and reduced levels of proinflammatory cytokines (TNFα, IL1β and IL-8). Therefore,the investigators believe that the "beneficial" bacteria from Visbiome will accelerate the normalization of gut immune cells and function in HIV-infected INRs. It is hypothesized consumption of Visbiome for 48 weeks will help restore the immune system in INRs who have suboptimal immune reconstitution to currently available ART. Resolution of gut immune cells will mean that microbial translocation and immune activation will be normalized and will reduce the rates of HIV-associated comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Male adult (age >18 years)
* Currently on ART (>2 years but <10 years)
* Undetectable HIV-1 viral load <50 copies/ml for the past 2 years (1 viral blip below 500 copies/ml permitted in the past year)
* Last CD4 count <350 cells/μl, and >70% over the past 2 years <350 cells/μl
* Ability to provide informed consent

Exclusion Criteria:

* Current alcohol or substance use judged by the Investigator to potentially interfere with subject study compliance
* Taking pharmaceutical-grade probiotics
* Any of the following abnormal laboratory results in screening:

  * Hemoglobin <85 g/L
  * Neutrophil count <750 cells/μl
  * Platelet count <50,000 cells/μL
  * AST or ALT >5X the upper limit of normal
* Colitis
* Liver fibrosis (decompensated cirrhosis), portal hypertension or clinical hepatitis
* Other significant underlying disease (non-HIV-1) that might impinge upon disease progression or death

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Percent change in blood immune activation | 48 weeks
  Percent change in blood immune activation (co-expression of CD38 and HLA-DR) on CD8 T cells at week 48 in participants randomized to probiotic Visbiome versus the placebo arm

SECONDARY OUTCOMES:
Level of microbial translocation (including LSP and sCD14) | 48 weeks
Plasma level of inflammation and coagulation (including IL-6, D-dimer and CRP) | 48 weeks
Number and function of gut immune cells (including CD4 T cell subsets) | 48 weeks
Intestinal permeability (Lac/Mac ratio) | 48 weeks
Bacterial community diversity, determined by 16s rRNA gene sequencing of penile swabs | 48 weeks
Bacterial community composition, determined by 16s rRNA gene sequencing of penile swabs | 48 weeks
Gut HIV DNA levels | 48 weeks
Canadian Diet History Questionnaire | 48 weeks
Safety assessed by AE monitoring and participant questionnaire | 48 weeks
Tolerability of Visbiome assessed by AE monitoring and participant questionnaire | 48 weeks
Adherence to Visbiome assessed by participant questionnaire and sachet count | 48 weeks

OTHER OUTCOMES:
Metabolomic measurements: vitamin D levels, glucose measurements, insulin levels and lipid profiling | 48 weeks
Microbiome analysis by 16s rRNA bacterial DNA isolated from penile swabs | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Kaul, MD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Maple Leaf Medical Clinic, Toronto, Ontario
  - Toronto General Hospital, UHN, Toronto, Ontario

REFERENCES:
- [Derived] Rousseau RK, Walmsley SL, Lee T, Rosenes R, Reinhard RJ, Malazogu F, Benko E, Huibner S, Kovacs CM, Singer J, Kim CJ, Kaul R. Randomized, Blinded, Placebo-Controlled Trial of De Simone Formulation Probiotic During HIV-Associated Suboptimal CD4+ T Cell Recovery. J Acquir Immune Defic Syndr. 2022 Feb 1;89(2):199-207. doi: 10.1097/QAI.0000000000002840. PMID 34693932